CLINICAL TRIAL: NCT07020143
Title: Chinese University Students' Death Attitudes and Their Initial Sandplay Characteristics
Status: Not yet recruiting | Type: Observational
Sponsor: Kai Huang (Other)
Responsible Party: Sponsor-Investigator, Kai Huang, Assistant Professor, Ocean University of China
Organization: Ocean University of China (Other)
Other Study IDs: OUCPHECC2025032202
Record Dates: First submitted 2025-05-15; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Death Attitude (Implicit/Explicit); Sandplay Therapy
Keywords: Chinese university students; implicit and explicit attitudes; death attitudes; the characteristics of initial sandplay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese university students: The study firstly explored the correlation between the implicit death attitudes and the explicit death attitudes by making pearson product-difference correlation between the implicit effect value D-value of the SC-IAT and the mean value of the sub-dimensions of the DAP-R. Secondly, based on the DAP-R scores, the university students with external death attitudes were categorized into positive and negative groups; based on the D values of the implicit effects of the SC-IAT, the university students with internal death attitudes were categorized into positive and negative groups, and the significance of the differences was investigated by conducting independent sample t-tests on the initial sandplay characteristics of the university students of the two groups respectively.

SUMMARY:
Death attitudes are different emotional reactions, evaluations, and behavioral tendencies of individuals experiencing near-death or death scenes, including positive or negative attitudes toward death such as denial, fear, curiosity, acceptance, avoidance, anxiety, etc. Wilson proposed a dual-attitude model to differentiate between implicit death attitudes and explicit death attitudes. Subsequently, some scholars have launched a discussion on the measurement and validity of implicit attitudes, Schimmack reviewed the evidence and found that the validity of implicit attitudes was lower than that of explicit instruments in all domains, but could be used as a complementary measure of sensitive attitudes; there are also several studies suggesting that implicit attitudes toward death could play a complementary role in the assessment of suicidal risk, and Wong found that a color image-based implicit association test was superior to a text-based one.

Sandplay therapy was developed by Swiss psychologist Dore M. Kalff in 1954 by combining Jung's analytical psychology and projection techniques with Lowenfeld's "The world technique". It was introduced to Japan by Hayao Kawai, a Japanese clinical psychologist, and introduced to China by Risheng Zhang in 1998. Sandplay therapy as a kind of deep-level expressive art therapy that uses sandboxes and tools to work with the self of individual cases, inherits the theories of Jungian psychotherapy about interpretation and metaphorical symbols, and can help individual cases to present unconscious contents and accomplish certain organization and transformation, which is very helpful to the development of the unconscious. It has a theoretical basis for reflecting the individual's implicit attitude toward death. Sandplay can express deeper emotional contents through metaphors and symbols .

Initial sandplay is the first one or two sandplays produced by a case. Research on the characteristics of the initial sandplay is helpful for clinicians to better grasp the psychological state and psychological traits of similar groups of people . Risheng Zhang does not advocate for the use of sandplay as a diagnostic tool, but sandplay does have a certain degree of diagnostic function, and by comparing the characteristics with those of the normative group, it can be used as one of the bases for preliminary judgment of the visitor. Renhui Lv suggested that Kalf and subsequent different scholars have combined their own experience in clinical practice to summarize the different methods and concerns of the box court assessment, although subjective assessment is criticized by scholars who hold a scientistic viewpoint, but it has to be admitted that any objectivization means cannot replace the flexibility and wholeness of the subjective assessment. The analytical dimensions of this study were defined in conjunction with the analytical dimensions used by several researchers regarding the study of sandplay characteristics.

This study planned to recruit 100 subjects through double-blind randomization, from which at least 82 subjects were selected from university students who had no religious beliefs, had an age range of 20±2 years old, had normal vision or corrected vision, none of them had participated in similar experiments before, and were familiar with basic computer operations. The study was based on a two-dimensional model of death attitudes, i.e., death attitudes were categorized into exoteric and implicit attitudes, and exoteric death attitudes were measured using the Depiction of Attitudes Toward Death Scale-Revised (DAP-R), and implicit death attitudes were measured using the Single-Category Implicit Association Test (SC-IAT), respectively. The study first explored the correlation between implicit and explicit attitudes toward death by correlating the implicit effect value D of the SC-IAT with the mean of the subdimensions of the DAP-R as pearson product difference. Secondly, based on the DAP-R scores, the university students with external death attitudes were categorized into positive and negative groups; based on the D values of the implicit effects of the SC-IAT, the university students with internal death attitudes were categorized into positive and negative groups, and the significance of the differences was investigated by conducting independent samples t-tests on the box characteristics of the university students of the two groups respectively.

ELIGIBILITY:
Inclusion Criteria Be aged 18-22 years (20 ± 2 years old) Self-identified as Han Chinese ethnicity Currently enrolled as an undergraduate student Normal or corrected-to-normal vision No prior participation in similar psychological experiments (e.g., IAT, sandplay therapy) Proficient in basic computer operations (e.g., keyboard use, mouse navigation) Willing to provide written informed consent Exclusion Criteria Presence of diagnosed psychiatric disorders (e.g., major depressive disorder, PTSD) Regular use of psychotropic medications within the past 6 months Religious affiliation or spiritual practices influencing death-related beliefs History of traumatic bereavement (e.g., loss of immediate family member within 1 year) Physical disabilities affecting sandplay manipulation (e.g., severe hand tremor)

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The trial randomly and double-blindly recruited 100 Han Chinese, with no religious beliefs, age range of 20 ± 2 years old, university students to participate in the trial, the subjects had normal vision or corrected vision, none of them had previously participated in similar experiments, and they were familiar with basic computer operation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Sandplay Feature Profile (SFP) via Sandplay Therapy Observation Scale | 1 day
  Quantitative analysis of initial sandplay characteristics using 5 validated dimensions:
  Toy Utilization Index: Count of distinct categories used (person/animal/plant/etc.) Sand Manipulation Score: 0-3 scale (0=no manipulation; 3=landform creation) Construction Time: Minutes from first toy selection to completion Self-Representation Coding: 0-2 nominal scale (0=absent; 1=symbolic; 2=literal) Spatial Occupancy Ratio: Calculated as (used area/total sandbox area)×100%

SECONDARY OUTCOMES:
Death Attitude Implicit Association (DA-IA) via SC-IAT | 1 day
  Description: D-value computed using Greenwald's improved algorithm (2003), reflecting response time differences between compatible (death-negative association) and incompatible (death-positive association) trials

OTHER OUTCOMES:
Explicit Death Attitude Profile via DAP-R | 1 day
  Composite scores from Chinese-validated Death Attitude Profile-Revised:
  Negative Attitude Score: Sum of Fear (5 items) & Avoidance (7 items) subscales Positive Attitude Score: Sum of Neutral/Acceptance/Escape Acceptance subscales

CONTACTS AND LOCATIONS:
Locations (1):
- Ocean University of China, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided